CLINICAL TRIAL: NCT04989309
Title: The Role of Frontal and Temporal Brain Areas in the Perception of Phonetic Category Structure
Brief Title: Left and Right Hemisphere Contributions to Speech Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Emily Myers, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H21-0046; R01DC013064 (NIH)
Record Dates: First submitted 2021-07-06; First posted 2021-08-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-12

CONDITIONS: Neural Bases of Speech Perception
Keywords: Speech perception; Left temporal lobe; Right temporal lobe
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will receive blocks of stimulation at the left temporal lobe, right temporal lobe, and vertex, with the order of stimulation counterbalanced across participants (a crossover design). All analysis is within-subject.
  Participants in each arm will hear different types of speech stimuli, which allows for the assessment of the effect of stimulation at different stimulation sites on processing that specific aspect of the speech signal.
Who Masked: Participant
Masking Description: Participants will receive stimulation at different sites (left and right temporal areas, vertex control), and may be aware of the location of placement of the TMS coil, so in a strict sense participants cannot be fully unaware of the stimulation site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experiment 2. Phonetic precision disrupted by TMS (Experimental): Experiment 2 tests the influence of temporary disruption of activity within the left or right temporal cortex on the speed and precision of phonetic decisions compared to vertex stimulation. Participants will receive stimulation at all three sites (left temporal, right temporal, vertex, with order of stimulation counterbalanced across participants). Immediately following stimulation pulses, participants will perform a visual analog scale (VAS) phonetic rating task on tokens from the four continua, embedded in speech-shaped noise. To control for the possibility that TMS leads to a generalized deficit in categorization, a control task will involve categorization of visual objects on a morphed "dog" to "cat" object continuum. (We expect this task to be unaffected by TMS). The variables of interest are the steepness of the categorization curve, mean reaction time to all items on the continuum, and the difference in reaction time for boundary vs. endpoint tokens.
  Interventions: Device: Transcranial Magnetic Stimulation
- Experiment 3. Phonetic ambiguity in continuous speech (Experimental): Experiment 3 is designed to test whether left vs. right temporal lobe stimulation selectively disrupts processing of naturally-occurring phonetic ambiguity as compared to vertex stimulation (control). Participants will receive stimulation at all three sites (left temporal, right temporal, vertex, with order of stimulation counterbalanced across participants). Stimuli will be nonsense sentences produced clearly or in a casual register. By-sentence phonetic ambiguity is estimated by the proximity of each token to other vowels belonging to different categories. Sentences will be embedded in speech-shaped noise to increase difficulty. Participants will listen to each sentence, then respond whether a visually-presented probe word appeared in the sentence ("BRASS?"). Dependent variables are accuracy and reaction time on this probe verification task.
  Interventions: Device: Transcranial Magnetic Stimulation
- Experiment 6: Disruption of talker-specific phonetic learning using TMS. (Experimental): Experiment 6 is designed to test whether disruption of activity in left or right temporal regions (vs. vertex control) using TMS interferes with talker-specific learning. Participants will receive stimulation at all three sites (left temporal, right temporal, vertex, with order of stimulation counterbalanced across participants). The study uses a training paradigm where one talker's speech is manipulated to always have relatively short voice onset times (VOTs) for voiceless stops (e.g., /k/ in "coal") and another to have relatively long VOTs. Immediately after stimulation, listeners will undergo a training trial where they identify sounds as mapping to Talker 1 or Talker 2's voice, and to the word (e.g. "gain" vs. "cane"). At test, listeners hear two VOT variants and are asked which is more typical of that talker's speech. The dependent variable is the accuracy of reporting which variant is typical of the talker.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS will be delivered in 10 Hz pulses for 2.5 seconds, with behavioral measures of speech perception and object categorization immediately following each pulse. TMS at this schedule is thought to temporarily disrupt activity at the stimulation site.

SUMMARY:
Left and right temporal brain areas are thought to contribute to speech perception, but the division of labor between left and right hemisphere regions is still unclear. Here we use transcranial magnetic stimulation (TMS) to stimulate left and right temporal foci and a vertex control site to temporarily disrupt activation at the stimulation site, using a "virtual lesion" approach to test the effect of stimulation site on a series of speech perception tasks.

This portion of the project is basic research. However, since TMS is viewed as an intervention, studies involving TMS in this grant are considered clinical trials.

DETAILED DESCRIPTION:
This study uses TMS to temporarily disrupt neural activity in the left and right temporal cortex and examine the effect of this disruption on speech perception tasks. Vertex stimulation is included as a control condition against which left and right superior temporal stimulation effects are compared. Adult participants first undergo structural MRI and a speech localizer using functional MRI to identify speech-sensitive voxels in the left and right temporal cortex. These regions are set by-participant as the foci for stimulation. Stimulation site is blocked, and typically distributed across sessions. 10 Hz pulse trains of 2.5 sec each are delivered to the stimulation site, with an auditory stimulus arriving either immediately after the last pulse (Exps 2 and 6) or, for longer sentence level stimuli (Exp 3), during the pulse train. Behavioral measures include accuracy and reaction times to rate phonetic stimuli (Exp 2), detect the presence of a probe word in the preceding sentence (Exp 3), or categorize stimuli by phonetic contrast and talker (Exp 6).

ELIGIBILITY:
Inclusion Criteria:

* Monolingual native speaker of English
* No history of neurological impairments or disease
* Free of speech and language disorders (per self-report, and confirmed by short language battery described by Fidler, Vance, & Plante, 2011)
* Pure-tone thresholds of 30 decibels or better in both ears (no worse than mild hearing loss), with no more than 15 dB between-ear difference.
* Right-handed, as confirmed by Oldfield Handedness Inventory

Exclusion Criteria:

* Any condition where TMS would be contraindicated according to the most recent guidelines, including, but not limited to:

  * History of seizure or epilepsy
  * Metal in the skull
  * Use of legal or illicit drugs that can potentially reduce the threshold for seizure. As examples, we list some exclusionary drugs in each of the following categories. This is not an exhaustive list of the exclusionary drugs. We consult with faculty in the University of Connecticut College of Pharmacy to check for seizure risk with other drugs that participants report.

    * Antidepressants including Imipramine, amitriptyline, sertraline, venlafaxine, buproprion
    * Antipsychotics including Chlorpromazine, clozapine, haloperidol, aripiprazole
    * Antivirals including foscarnet, ganciclovir
    * Antiparasitics including chloroquine, mefloquine (antiparasitics)
    * Antibiotics including penicillin, ampicillin
    * Immunosuppressants including cyclosporin
    * Anticholinergenics
    * Antihistimines (including over-the-counter drugs like Claritin & Benadryl)
    * Sympathomimetics (including Sudafed, Ritalin).
    * Illegal drugs such as methamphetamines, cocaine, MDMA, ketamine.
  * Diagnosis of a psychiatric disorder (per self-report)
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Categorization accuracy | Immediately following the stimulation pulses (within one second of the final pulse).
  Participants categorize items which vary along a perceptual continuum. Steepness of the categorization curve is extracted to estimate categorization accuracy.
Two-alternative forced choice accuracy | Immediately following the stimulation pulses (within one second of the final pulse).
  Participants are given two options and asked to indicate which item they heard in the previous signal. Accuracy in making this decision is a primary outcome measure.
Two-alternative forced choice reaction time | Immediately following the stimulation pulses (within one second of the final pulse).
  Participants are given two options and asked to indicate which item they heard in the previous signal. Reaction time to make this decision is a primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of these studies will be used for teaching, research publications, and presentation at scientific meetings. De-identified raw data of all types (behavioral, MRI) will be available upon request after publication. MRI data will be processed ("skull stripped") to remove any identifiable anatomy before archival. We will archive data locally using Brain Imaging Data Structure (BIDS) naming conventions to facilitate data sharing.
  We plan to pre-register behavioral studies on the Open Science Framework (or similar platforms), and in the interests of scientific transparency, we will post de-identified behavioral data and analysis code on Open Science Framework or GitHub.
Supporting Information: SAP, Analytic Code
Time Frame: We will share data and code upon publication, and de-identified data will be available indefinitely.
Access Criteria: Open

REFERENCES:
- [Background] Kennedy-Higgins D, Devlin JT, Nuttall HE, Adank P. The Causal Role of Left and Right Superior Temporal Gyri in Speech Perception in Noise: A Transcranial Magnetic Stimulation Study. J Cogn Neurosci. 2020 Jun;32(6):1092-1103. doi: 10.1162/jocn_a_01521. Epub 2020 Jan 14. PMID 31933438
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615